CLINICAL TRIAL: NCT00904527
Title: Interest of Relaxation From Patients With Pain Due to Migraine
Acronym: MIGREL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0601001b
Record Dates: First submitted 2009-05-18; First posted 2009-05-19 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Migraine
Keywords: Relaxation (Schultz); Migraine; antipain center
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Relaxation (Experimental): Relaxation (Schultz)+ medical treatment (beta-bloquant or Oxetorone)+ patient's education
  Interventions: Behavioral: relaxation (Schultz)
- without relaxation (No Intervention): Patients have no relaxation (only medical treatment+ education)

INTERVENTIONS:
Behavioral: relaxation (Schultz) — Patients have relaxation consultations during 2 months
  Arms: Relaxation

SUMMARY:
The purpose of this study is to determine whether relaxation (autogenic training of Schultz) is effective in treatment for migraine.

DETAILED DESCRIPTION:
This randomized, multicenter study compares 2 parallel groups of patients with migraine :

* I: patients are treated with relaxation + medical treatment (beta-bloquant or Oxetorone)+ patients' education
* II: patients are treated only with medical treatment + patients' education.

Visit 1 : 1 month before randomization for patient's selection and baseline data

Visit 2 (J0): inclusion (randomization) During the first 2 months patients from group I benefit from relaxation consultations.

Visit 3 (2 months after randomization)and visit 4 (4 months after randomization) : evaluation of the efficacy of the two treatment strategies.

Primary endpoint :

- number of days with migraine per month from J0 to visit 4.

Secondary endpoints :

* monthly drug consumption
* percentage of patients who respond (50 % frequency reduction)
* quality of life (SF 36)

Each day, patients note in a notebook if a migraine appears and its intensity.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* 5 to 14 days of migraines per month

Exclusion Criteria:

* Headache by medication abuse
* Patients who already know relaxation technics
* Depression
* Contra indication of using beta-bloquant or Oxetorone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-06; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Comparison of reduction of migraine frequency between the 2 groups (with or without relaxation) | 4 months

SECONDARY OUTCOMES:
Comparison between the 2 groups of intensity of migraine, medication use and quality of life | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: LAURENT Bernard, MD PhD, Study Director — Centre Hospitalier Universitaire de Saint Etienne; PICKERING Gisèle, MD, Study Chair — Centre d'Investigation Clinique de Clermont-Ferrand
Locations (9):
- France (9):
  - Consultation de la douleur du CHU d'Amiens, Amiens
  - UTCD - CHU Pellegrin, Bordeaux
  - CETD - CHU de Caen, Caen
  - CETD du CHU Gabriel Montpied, Clermont-Ferrand
  - CETD CHU de Grenoble, Grenoble
  - Consultation de la douleur - CH Emile Roux, Le Puy-en-Velay
  - CETD CH de Nemours, Nemours
  - CETD du CHU de Saint-ETienne, Saint-Etienne
  - CETD Hôpital Rangueil, Toulouse